CLINICAL TRIAL: NCT01882205
Title: Endoscopic Screening for Dysplasia in Patients With Longstanding Ulcerative Colitis: Classical Chromo-endoscopy Versus NBI , FICE and EPK-i.
Brief Title: Comparison Between Chromoendoscopy and Virtual Chromoendoscopy (NBI, I-scan, FICE) for Detection of Neoplasia in Long Standing Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: H.-Hartziekenhuis Roeselare-Menen VZW, Belgium. (Unknown); McGill University (Other); Maastricht University Medical Center (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S50565
Record Dates: First submitted 2013-06-12; First posted 2013-06-20 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; DALM; chromoendoscopy; dysplasia; virtual chromoendoscopy; FICE; NBI; I-scan
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- OLYMPUS CHROMO (Active Comparator): Group A: HDTV Olympus colonoscopes and Chromo-endoscopy, methylene blue 0.1%
  Interventions: Procedure: Chromoendoscopy
- OLYMPUS NBI (Experimental): Group B: Virtual chromoendoscopy: HDTV Olympus colonoscopes and Narrow band Imaging (NBI)
  Interventions: Device: Virtual chromoendoscopy
- FUJINON CHROMO (Active Comparator): Group C: CCD Fujinon colonoscopes and Chromo-endoscopy, methylene blue 0.1%
  Interventions: Procedure: Chromoendoscopy
- FUJINON FICE (Experimental): Group D: Virtual chromoendoscopy: CCD Fujinon colonoscopes and Fujinon Intelligent Color Enhancement n° 4
  Interventions: Device: Virtual chromoendoscopy
- PENTAX CHROMO (Active Comparator): Group E: HD-Pentax colonoscopes and Chromo-endoscopy, methylene blue 0.1%
  Interventions: Procedure: Chromoendoscopy
- PENTX i-scan (Experimental): Group F: Virtual chromoendoscopy: HD Pentax colonoscopes and I-scan 2 settings
  Interventions: Device: Virtual chromoendoscopy

INTERVENTIONS:
Device: Virtual chromoendoscopy
  Other Names: Narrow band Imaging (NBI); Fujinon Intelligent Color Enhancement; I-scan
  Arms: FUJINON FICE; OLYMPUS NBI; PENTX i-scan
Procedure: Chromoendoscopy — Panchromocolonoscopy with methyleen blue 0.1%
  Arms: FUJINON CHROMO; OLYMPUS CHROMO; PENTAX CHROMO

SUMMARY:
The risk for colon cancer in patients with longstanding ulcerative colitis exceeding the rectum is increased and therefore patients should be enrolled in a surveillance program eight years after the diagnosis. Until today, official international guidelines for endoscopic screening in patients with ulcerative colitis advise to take 4 biopsies every 10 centimeters (with a minimum of 32) and of each suspected visible lesion. These guidelines are merely based on consensus during expert opinion meetings rather than evidence based. Recent studies have shown that chromo-endoscopy guided biopsies significantly reduced the number of biopsies for each procedure and detected more neoplastic lesions. Chromo-endoscopy is therefore considered the gold standard in this study in which we want to compare it to the performance and efficiency of new endoscopic imaging techniques.

Narrow-Band Imaging (NBI) selectively uses certain wavelengths of the visible light leading to a shift in the excitation spectrum towards blue light. The first studies with NBI showed that the additional value of NBI in the detection of neoplastic lesions is comparable to chromo-endoscopy, but time saving and easier to perform. The Fujinon Intelligent Chromo-Endoscopy (FICE) system uses a similar theoretical principal as NBI but this is achieved via the use of post hoc computer algorithms, applying different filters to the stored endoscopic images and enabling a theoretically endless number of combinations of filters that can be used. The Pentax I-scan system also allows post hoc modification of the images. On the one hand, surface enhancement enables to better highlight mucosal changes. Spectral modification allows to apply different modes in analogy with to FICE system.

These new imaging techniques have a theoretical advantage which is extendedly used for sales purposes but has however so far not been proven in ulcerative colitis patients. We want to test their clinical use in the screening for neoplastic lesions in patients with long standing ulcerative colitis.

DETAILED DESCRIPTION:
The risk for colon cancer in patients with longstanding ulcerative colitis exceeding the rectum is increased and therefore patients should be enrolled in a surveillance program eight years after the diagnosis. Surveillance endoscopies are advised 8 to 10 years after the diagnosis of ulcerative colitis. The first decade every 3 years, the second decade every 2 years and thereafter every year Until today, most official international guidelines for endoscopic screening in patients with ulcerative colitis advise to take 4 random biopsies every 10 centimeters (with a minimum of 32) and of each suspected visible lesion using standard white light endoscopy.

These guidelines are merely based on consensus during expert opinion meetings rather than evidence based.

However, some studies have shown that the sensitivity for the detection of dysplasia during colonoscopy in patients with ulcerative colitis can significantly be enhanced by using chromo-endoscopy. These studies used methylene blue or indigo carmine as a contrast agent with or without high magnification endoscopy. Chromo-endoscopy guided targeted biopsies significantly reduced the number of biopsies for each procedure and detected more neoplastic lesions. It was therefore concluded that colonoscopy with chromo-endoscopy guided biopsies is more efficient and cost saving. Chromo-endoscopy with targeted biopsies is an alternative to white light endoscopy with random biopsies every 10cm. The European Crohn and Colitis association now suggests that the use of methylene blue or indigo carmine chromoendoscopy is an alternative to random biopsies for appropriately trained endoscopists and is superior to random biopsies in the detection rate of neoplastic lesions In this study we want to compare chromoendoscopy with targeted biopsies as the gold standard with new new endoscopic image techniques called virtual chromoendoscopy.

From 2005 new endoscopic imaging modalities have been commercialized and are now generally available to gastroenterologists. They all claim a theoretical advantage in comparison to standard white light high resolution video endoscopy. These new techniques are called virtual chromoendoscopy (VC). There are three different systems developed by the three major competitors of endoscopic equipment: Olympus, Pentax and Fujinon.

Narrow-Band Imaging (NBI) is developed by Olympus inc. and selectively uses certain wavelengths of the visible light leading to a shift in the excitation spectrum towards blue light. The intensity of the blue bandwidth is also enhanced. This leads to a more superficial penetration of the emitted light into the mucosa of the intestine and enhancement of more superficial structures (e.g. irregularities, small flat lesions or polyps) and small superficial mucosal vessels (indicative of neoplasia).

The first studies using NBI in Barrett's esophagus demonstrated that the additional value of NBI in the detection of neoplastic lesions is comparable to chromo-endoscopy (Kara et al., 2005). However NBI is time saving and easier to perform than chromo-endoscopy because there is no need to additionally spray dye onto the mucosa.

In a standard population screening study, NBI has shown to aid in the detection and characterization of polyps in the colon. In particular the presence of a brownish meshed capillary network has a high diagnostic value in the prediction of the neoplastic nature of a lesion.

In a very recent tandem study in which white light endoscopy was compared with NBI in 48 patients with longstanding UC there was no additional benefit of NBI. In the 25 patients who were first endoscoped with white light 8 dysplastic lesions were found. After NBI imaging another 7 lesions were found. In the 23 patients which were first imaged with NBI 7 lesions were found and an additional 8 after white light endoscopy (Van den Broek FJ et al 2011.

The Fujinon Intelligent Chromo-Endoscopy (FICE) system uses a similar theoretical principal as NBI but this is achieved via the use of post hoc computer algorithms, applying different filters to the stored endoscopic images and enabling a theoretically endless number of combinations of filters that can be used. Currently 10 different spectrum filters can be used. There are predefined settings for visualization of the colonic mucosa. There are no previous data comparing white light endoscopy and FICE in the detection of dysplasia in longstanding ulcerative colitis.

Finally, Pentax released a new high definition endoscopy system in 2007, the I-scan system, which also allows post hoc modification of the images. On the one hand, surface enhancement enables to better highlight mucosal changes. Spectral modification allows to apply different modes in analogy with to FICE system. For instance the p-mode for pattern recognition helps to accentuate epithelial features. The TE-mode helps to assess the vasculature of the gastrointestinal mucosa. Recently new filters were developed such as the colon mode, specifically designed for the colon. In one study VC with I-scan TE-mode was compared to CE and standard white light endoscopy in 69 patients. In both the VC and CE mode 11 dysplastic lesions were found (Hoffman et al 2010). Data about the improvement of detection of dysplasia are lacking until now.

Adjustment of the light spectrum is usually combined with a better and higher image resolution of the new generation endoscopes. Fujinon and Pentax use a so called super-CCD to increase the pixel resolution of the scope to 1.300.000 and 1.400.000 respectively and combined it with a DVI output signal. Olympus opted for an improved video resolution by incorporating high definition television (HDTV) in the latest processors.

These new imaging techniques have a theoretical advantage which is extendedly used for sales purposes but has however so far not been proven in ulcerative colitis patients. We want to test their clinical use in the screening for neoplastic lesions in patients with long standing ulcerative colitis. The scientific and clinical relevance of this study is clear. If NBI and/or FICE and/or I-scan have a better detection rate than chromo-endoscopy, the latter can be replaced by virtual chromo-endoscopy. Even if the detection by NBI and/or FICE and/or I-scan is not statistically different from standard chromo-endoscopy, they still can replace the latter because it is technically easier to use. If however these techniques have a lower adenoma detection rate than classical chromo-endoscopy we will be able to show that there is no place for these techniques in the detection of UC related neoplasia, despite the theoretical advantage.

Because the multicenter character of the study, and the availability of only one system in most hospitals, we will test the differences between all three modalities and classical chromoendodoscopy.

The endoscopic procedure as such is not much different from a standard endoscopic procedure that patient should be advised to undergo according to good clinical practice. The bowel preparation is similar as in a normal colonoscopy, and can be performed either at home or in the endoscopy department. The endoscopes used in the study include the H180Q series of Olympus, the 5000 series of Fujinon and the HD series of Pentax. They are not different in terms of design or size compared to standard colonoscopies and are all commercially available.

Patients will be randomized between one of the following techniques:

1. Chromo-endoscopy with methylene blue 0,1% (groups A-C-E) An Olympus spray catheter is used through the biopsy channel of the endoscope to apply the dye, a saline solution with methylene blue in a concentration of 0.1%. This technique was already validated in previous studies. Besides the extra time needed for dying the entire colon mucosa, no other manipulations are needed for this technique. Moreover, the time needed to dye can be recovered because only chromo-endoscopy guided biopsies will be taken instead of random biopsies throughout the colon, which normally also requires a considerable amount of time. Previous studies using chromo-endoscopy versus conventional screening colonoscopy did not show a significant difference in total procedure time. The endoscopes used do not differ from the ones used in the other randomization arms and include either an Olympus H180Q colonoscope, Fujinon EC 590 ZW/M colonoscope or a Pentax 3890i colonoscope. All three endoscopes are CE approved and are commercially available.
2. Narrow band imaging with HDTV (Group B) This technique involves an Olympus H180Q colonoscope that is CE approved and commercially available. The procedure involves a normal white light endoscopy during progression of the scope. Once the caecum is reached the entire procedure will be performed in NBI modus. This has no influence or side effects for the patients because NBI modus is switched on by pushing a button on the scope.
3. Fujinon Intelligent Color Enhancement (FICE) with super CCD chip (Group D) This technique involves a Fujinon EC 590ZW/M colonoscope that is CE approved and commercially available. The procedure involves a normal white light endoscopy during progression of the scope. Once the caecum is reached the entire procedure will be performed in FICE modus n° 4. This has no influence or side effects for the patients because FICE modus is switched on by pushing a button on the scope.
4. I-scan with High Definition colonoscope (group F) This technique involves a PENTAX EC3890Fi colonoscope that is CE approved and commercially available. The procedure involves a normal white light endoscopy during progression of the scope. Once the caecum is reached the entire procedure will be performed in the TE- modus (Tissue enhancement mode) with surface enhancement on medium (range low-medium-high). This has no influence or side effects for the patients because the c- modus is switched on by pushing a button on the scope.

Only targeted biopsies of visible mucosal abnormalities during chromo-endoscopy, NBI, FICE or I-scan endoscopy will be taken. This is in concordance with the standard approach during chromo-endoscopy directed screening colonoscopy for ulcerative colitis. The disposable biopsy forceps are commercially available (Boston Scientific) and do not differ from the ones used during normal endoscopic procedures.

Power calculation

A power analysis was performed to detect a statistical significance between group A and B, group C and D and between group E and F. In a previous study dysplasia was found three times more often using CE compared to white light endoscopy: 32/84 versus 10/81 patients. This wil give an increase from approximate 10 to 30 percent. It is expected that in both study groups the percentage of dysplasia equals.

Inclusion of 67 patients in each group will allow to detect a 20% increase of dysplasia from 10 to 30% compared to white light endoscopy with a power of 80% (beta error 0.2; alpha error 0.05). We expect to include a total of (67 x 6 =) 402 patients in the study.

5.5 Co-variables

Multiple factors will be used as co-variables

* Age
* Duration of disease
* Existence of PSC
* Use of medication

  * Mesalazine/Sulfazalazine
  * Thiopurines
  * Biologicals

ELIGIBILITY:
Inclusion Criteria:

* Patients with longstanding ulcerative colitis ( 8 years after diagnosis or pancolitis and 10 years after diagnosis of left-sided colitis)
* Signed informed consent form
* Previous surveillance endoscopy > 1 year

Exclusion Criteria:

* Active ulcerative colitis, > 20 cm from the margo ani
* Personal history of colorectal cancer
* Allergy or intolerance to methylene blue
* Refusing or incapable to agree with informed consent
* Age younger than 18 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2008-05; Primary Completion 2018-12 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The difference in total number of neoplastic lesions detected by chromoendoscopy and virtual chromoendoscopy | The primary endpoint can be assessed when pathology results are available : 2 weeks after endoscopy
  The primary endpoint will be assessed in three subgroups comparing :
  1 )Group A: HDTV Olympus colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group B: HDTV Olympus colonoscopes and Narrow band Imaging (NBI)
  2) Group C: CCD Fujinon colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group D: CCD Fujinon colonoscopes and Fujinon Intelligent Color Enhancement
  3) Group E: HD-Pentax colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group F: HD Pentax colonoscopes and I-scan
  As such this is not a comparison between different endoscopy systems, but a comparison of chromoendoscopy and virtual chromoendoscopy within each different system.

SECONDARY OUTCOMES:
Duration of total endoscopic procedure time and of endoscopic procedure time during retraction for each technique. | The endpoint can be assessed immediately after the endoscopy.
  The total endoscopy time is recorded from the start until the end of the entire procedure. After the caecum is reached, time is recorded. Total retraction time is the time between reaching the caecum and the end of the procedure and includes time for rinsing, dye spraying, biopsy or poliepectomy.
The difference in neoplasia detection rate (i.e. the number of patients with at least one neoplastic lesion) between chromoendoscopy and virtual chromoendoscopy. | The endpoint can be assessed when pathology results are available : 2 weeks after endoscopy
  The endpoint will be assessed in three subgroups comparing :
  1 )Group A: HDTV Olympus colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group B: HDTV Olympus colonoscopes and Narrow band Imaging (NBI) 2) Group C: CCD Fujinon colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group D: CCD Fujinon colonoscopes and Fujinon Intelligent Color Enhancement 3) Group E: HD-Pentax colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group F: HD Pentax colonoscopes and I-scan As such this is not a comparison between different endoscopy systems, but a comparison of chromoendoscopy and virtual chromoendoscopy within each different system.
The difference in the ratio number of neoplastic lesions/ total number of lesions between chromoendoscopy and virtual chromoendoscopy | The endpoint can be assessed when pathology results are available : 2 weeks after endoscopy
  The endpoint will be assessed in three subgroups comparing :
  1 )Group A: HDTV Olympus colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group B: HDTV Olympus colonoscopes and Narrow band Imaging (NBI) 2) Group C: CCD Fujinon colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group D: CCD Fujinon colonoscopes and Fujinon Intelligent Color Enhancement 3) Group E: HD-Pentax colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group F: HD Pentax colonoscopes and I-scan As such this is not a comparison between different endoscopy systems, but a comparison of chromoendoscopy and virtual chromoendoscopy within each different system.

OTHER OUTCOMES:
The difference in total number of non-neoplastic lesions detected by chromoendoscopy and virtual chromoendoscopy | The endpoint can be assessed when pathology results are available : 2 weeks after endoscopy
  The endpoint will be assessed in three subgroups comparing :
  1 )Group A: HDTV Olympus colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group B: HDTV Olympus colonoscopes and Narrow band Imaging (NBI) 2) Group C: CCD Fujinon colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group D: CCD Fujinon colonoscopes and Fujinon Intelligent Color Enhancement 3) Group E: HD-Pentax colonoscopes and Chromo-endoscopy, methylene blue 0.1% to Group F: HD Pentax colonoscopes and I-scan As such this is not a comparison between different endoscopy systems, but a comparison of chromoendoscopy and virtual chromoendoscopy within each different system.
Number of biopsies per colonoscopy taken in the different groups. | Endpoint can be assessed immediately after endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Raf Bisschops, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (5):
- Belgium (2):
  - University Hospitals Leuven, Leuven
  - H.-Hartziekenhuis Roeselare-Menen VZW, Roeselaere
- McGill University Health Center, Montreal, Canada
- Copenhagen University Hospital Herlev, Copenhagen, Denmark
- Academic Medical center Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Bisschops R, Bessissow T, Dekker E, East JE, Para-Blanco A, Ragunath K, Bhandari P, Rutter M, Schoon E, Wilson A, John JM, Van Steen K, Baert F, Ferrante M. Pit pattern analysis with high-definition chromoendoscopy and narrow-band imaging for optical diagnosis of dysplasia in patients with ulcerative colitis. Gastrointest Endosc. 2017 Dec;86(6):1100-1106.e1. doi: 10.1016/j.gie.2017.09.024. Epub 2017 Oct 3. PMID 28986266
- [Derived] Bisschops R, Bessissow T, Joseph JA, Baert F, Ferrante M, Ballet V, Willekens H, Demedts I, Geboes K, De Hertogh G, Vermeire S, Rutgeerts P, Van Assche G. Chromoendoscopy versus narrow band imaging in UC: a prospective randomised controlled trial. Gut. 2018 Jun;67(6):1087-1094. doi: 10.1136/gutjnl-2016-313213. Epub 2017 Jul 11. PMID 28698230